CLINICAL TRIAL: NCT07080060
Title: Effects of Niel-Asher Technique Versus Spencer Technique Along With Conventional Therapy on Pain, Range of Motion, and Functional Status in Frozen Shoulder Patients
Brief Title: Comparison of Niel-Asher and Spencer Techniques in Frozen Shoulder Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0167- Minahil
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Frozen Shoulder; Adhesive Capsulitis
Keywords: Manual Therapy; Niel-Asher Technique; Spencer Technique; Pain; Range of motion
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niel-Asher Technique (Experimental): Participants in this group will receive the Niel-Asher Technique, a manual therapy approach focusing on trigger point release and myofascial decompression of the shoulder girdle. Treatment will involve structured pressure techniques applied to specific muscular trigger points including the infraspinatus, supraspinatus, subscapularis, and levator scapulae. The intervention will be delivered in side-lying and sitting positions.
  Interventions: Other: Niel-Asher Technique
- Spencer Technique (Experimental): Participants in this group will receive the Spencer Technique, an osteopathic manual therapy consisting of eight mobilization steps: extension, flexion, circumduction with compression, circumduction with distraction, abduction, adduction with external rotation, internal rotation, and traction stretch. Each movement will be performed with patient participation using muscle energy techniques.
  Interventions: Other: Spencer Technique

INTERVENTIONS:
Other: Niel-Asher Technique — Participants in this group will receive the Niel-Asher Technique, a manual therapy approach focusing on trigger point release and myofascial decompression of the shoulder girdle. Treatment will involve structured pressure techniques applied to specific muscular trigger points including the infraspinatus, supraspinatus, subscapularis, and levator scapulae. The intervention will be delivered in side-lying and sitting positions.
  Conventional physiotherapy, includes a 10-minute hot pack, 15-minute TENS, Codman exercises, finger ladder exercises (2-3 sets, 3-5 repetitions), and capsular stretching (20-30 sec hold, 2-4 repetitions). Sessions will be conducted 3 times per week for 4 weeks.
  Arms: Niel-Asher Technique
Other: Spencer Technique — Participants in this group will receive the Spencer Technique, an osteopathic manual therapy consisting of eight mobilization steps: extension, flexion, circumduction with compression, circumduction with distraction, abduction, adduction with external rotation, internal rotation, and traction stretch. Each movement will be performed with patient participation using muscle energy techniques.
  Conventional physiotherapy, includes a 10-minute hot pack, 15-minute TENS, Codman exercises, finger ladder exercises (2-3 sets, 3-5 repetitions), and capsular stretching (20-30 sec hold, 2-4 repetitions). Sessions will be conducted 3 times per week for 4 weeks.
  Arms: Spencer Technique

SUMMARY:
This study aims to compare the effectiveness of two manual therapy techniques-Niel-Asher Technique and Spencer Technique-when combined with conventional physiotherapy in treating patients with frozen shoulder (adhesive capsulitis). Frozen shoulder is a painful condition that limits movement and function of the shoulder joint. The study will include 44 adults aged 35 to 65 years who have been diagnosed with stage II frozen shoulder. Participants will be randomly assigned to one of two groups. Both groups will receive standard physiotherapy, including heat therapy, TENS, and stretching exercises. In addition, one group will receive the Niel-Asher Technique, while the other group will receive the Spencer Technique. Pain, range of motion, and shoulder function will be measured before and after a 4-week treatment period using validated tools such as the Visual Analogue Scale (VAS), a goniometer, and the Shoulder Pain and Disability Index (SPADI). The goal is to determine which manual therapy technique is more effective in improving symptoms and function in patients with frozen shoulder.

DETAILED DESCRIPTION:
Frozen shoulder, also known as adhesive capsulitis, is a common musculoskeletal condition characterised by pain, stiffness, and reduced range of motion of the glenohumeral joint. It is often associated with idiopathic onset, and can significantly impair daily activities and quality of life. While conventional physiotherapy-including modalities such as heat, TENS, and therapeutic exercise-forms the basis of treatment, there is growing evidence supporting the use of manual therapy techniques for enhanced outcomes.

This randomised controlled trial investigates the comparative effects of the Niel-Asher Technique and the Spencer Technique, each provided alongside standard conventional physiotherapy. A total of 44 patients meeting inclusion criteria (age 35-65 years, diagnosed with stage II adhesive capsulitis, and VAS pain score <7/10) will be enrolled and randomly assigned to one of two groups using computer-generated numbers and sealed envelope allocation.

Group A will receive the Niel-Asher Technique, which targets trigger points and myofascial release to reduce muscle guarding and pain. Group B will receive the Spencer Technique, a structured sequence of mobilisation techniques often used in osteopathic manual therapy. Both groups will also receive conventional therapy including moist heat, TENS, Codman exercises, finger ladder exercises, and capsular stretching.

The intervention will be administered three times per week over a 4-week period. Primary outcome measures include shoulder pain assessed by the Visual Analogue Scale (VAS), range of motion measured by a universal goniometer, and functional status assessed by the Shoulder Pain and Disability Index (SPADI).

Data will be analysed using SPSS 25.0. Parametric or non-parametric tests will be applied based on data distribution. The findings of this study aim to provide evidence for clinical decision-making in the manual therapy treatment of frozen shoulder and may help establish more effective, hands-on techniques in physiotherapy practice.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 35-65 years diagnosed with primary Adhesive Capsulitis.
* Both gender male and female.
* Both Active and passive Range of Motion is limited.
* Stage II Frozen Shoulder patients (Freezing Stage,3-9 months).
* More than 50% of range of motion is limited in Flexion, Abduction and External rotation as compared to unaffected side.
* Pain reported on VAS score <7/10 in shoulder region.
* Patients agree to sign written consent form.

Exclusion Criteria:

* Patients with systemic illness:
* Diabetes Mellitus, Thyroid disorders.
* Rheumatoid Arthritis, Malignancy.
* Patients with mechanical injuries like:
* Rotator Cuff injury, Ligamentous Injuries.23
* Previous Surgery or Manipulation under Anesthesia.
* Patients with Stage I, III, IV of Frozen Shoulder.
* Patient reported with VAS score >7/10 in shoulder region.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline and 4 Weeks Post-Treatment
  Pain intensity in the affected shoulder will be assessed using the Visual Analogue Scale (VAS), a validated 10-point scale where 0 indicates "no pain" and 10 indicates "worst imaginable pain." A decrease in score indicates pain reduction.
Shoulder Range of Motion (ROM) | Baseline and 4 Weeks Post-Treatment
  Shoulder joint range of motion, including flexion, abduction, and external rotation, will be measured using a universal goniometer. ROM will be recorded in degrees. An increase in ROM values indicates functional improvement.
Shoulder Pain and Disability Index (SPADI) | Baseline and 4 Weeks Post-Treatment
  Shoulder function will be evaluated using the Shoulder Pain and Disability Index (SPADI), a self-reported questionnaire assessing pain and disability. Scores range from 0 (no pain/disability) to 100 (maximum pain/disability). A reduction in score indicates functional improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Zia, Phd Scholar, Principal Investigator — Riphah International University/ Mayo Hospital
Locations (1):
- Noor Thalassemia Foundation, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavalleri E, Servadio A, Berardi A, Tofani M, Galeoto G. The effectiveness of physiotherapy in idiopathic or primary frozen shoulder. A systematic review and meta- analysis. MLTJ MUSCLES, LIGAMENTS AND TENDONS JOURNAL. 2020;10(1):24-39.
- [Background] Tang CK, Shih YF, Lee CS. The effect of muscle-biased manual therapy on shoulder kinematics, muscle performance, functional impairment, and pain in patients with frozen shoulder. J Hand Ther. 2025 Jan-Mar;38(1):42-51. doi: 10.1016/j.jht.2024.02.010. Epub 2024 Jun 29. PMID 38944638
- [Background] Raghav D, Krishnapandian PR, Dwivedi A. Comparative Effect of Niel-Asher Technique and Positional Release Technique on Pain, Active ROM and Functional Disability in Adhesive Capsulitis: An Experimental Study. JOURNAL OF CLINICAL AND DIAGNOSTIC RESEARCH. 2023 Apr 1;17(4):YC01-5.
- [Background] Phansopkar P, Qureshi MI. A Research Protocol on Comparative evaluation of Efficacy of Spencer Technique, Kaltenborn, Mulligan, and Maitland mobilization on Pain, Range of Motion and Functional Disability in Frozen Shoulder.
- [Background] Riaz H, Javed A, Ali H, Kazmi YA, Naz S, Javed Z. COMPARATIVE EFFECT OF SPENCER TECHNIQUE VS MULLIGAN MOBILIZATION ON ROM AND FUNCTIONAL DISABILITY AMONG ADHESIVE CAPSULITIS PATIENTS. Insights-Journal of Health and Rehabilitation. 2025 Jan 27;3(3 (Health & Rehab)):156-65.